CLINICAL TRIAL: NCT02235090
Title: Assessment of Feasibility and Statistical Reliability of Functional Outcomes Measurement in Neuromuscular Patients Without Trial Site Visiting by Standard Functional Scales and by Special Autonomic Device in Double-blind, Placebo Controlled Study of Cervical Spinal Cord Transdermal Direct Current Stimulation in Patients With Spinal Muscular Atrophy
Brief Title: Study of Feasibility to Reliably Measure Functional Abilities' Changes in Nonambulant Neuromuscular Patients Without Trial Site Visiting
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Trial was not started due to lack of funding and nobody received an intervention.
Sponsor: Charitable Foundation Children with Spinal Muscular Atrophy (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Other
Other Study IDs: CSMA-INPN-1
Record Dates: First submitted 2014-09-03; First posted 2014-09-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Spinal Muscular Atrophy; Neuromuscular Disorders
Keywords: Spinal muscular atrophy; Neuromuscular disorders; Outcome measures; Visit-free clinical trial design
MeSH Terms: conditions — Muscular Atrophy, Spinal; Neuromuscular Diseases

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- Zero-strength of direct current stimulation (Sham Comparator): Sham transdermal direct current stimulation of cervical spinal cord
  Interventions: Other: Direct current stimulation of cervical spinal cord
- 100 microamperes direct current stimulation (Experimental): Transdermal direct current stimulation of cervical spinal cord
  Interventions: Other: Direct current stimulation of cervical spinal cord
- 1 milliampere direct current stimulation (Experimental): Transdermal direct current stimulation of cervical spinal cord
  Interventions: Other: Direct current stimulation of cervical spinal cord

INTERVENTIONS:
Other: Direct current stimulation of cervical spinal cord — 10 minutes direct current stimulation of 0, 100 microamperes, 1 milliampere strengths applied through dermal electrodes to cervical spinal cord

SUMMARY:
Clinical trials organization in several neuromuscular disorders (NMD) has some specific issues. Nonambulant status and difficulties with transportation are among them. Moreover a lot of patients with NMD have so poor condition that even short transportation is able to worse it. Such situation forces researchers to limit a region of recruitment for clinical trials and to exclude from trials more severe subgroup of patients, which cause additional issues especially for rare diseases.

The purpose of this study is to prove hypothesis about possibility to reliably monitor patient condition remotely, without trial site visiting. Visit-free study design is potentially able to widen eligible patient population and to decrease patient dropout rate as well as burden of numerous assessments. Meanwhile assessment frequency could be increased enabling monitoring of short fluctuations in patients' condition.

Spinal muscular atrophy (SMA) is a rare neuromuscular condition to which all mentioned above issues are completely applicable. Direct current stimulation (DCS) of neural structures is well studied and safe intervention, however, its effects on SMA patients' strength and durability has not been reported for today. The investigators suppose that investigation of DCS action in SMA patient population is an adequate model for visit-free design feasibility, reliability and sensitivity evaluation.

ELIGIBILITY:
Inclusion Criteria:

* Signed informed consent
* 5q SMA confirmed by molecular testing

Exclusion Criteria:

* Need for ventilation
* Hypersensitivity (pain or allergic reaction) to current stimulation

Min Age: 5 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2016-10 (Actual); Primary Completion 2017-09-30 (Actual); Study Completion 2017-10-30 (Actual)

PRIMARY OUTCOMES:
Strength Changes from baseline measured by handheld myometry after spinal cord direct current stimulation of different intensity | Before and 0, 15, 30 minutes after spinal cord direct current stimulation

SECONDARY OUTCOMES:
Short time fluctuations of Hammersmith Functional Motor Scale indexes | Three times, three days consecutive measurement, every two months, assessed up to 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Andriy V. Shatillo, MD, PhD, Principal Investigator — State Institution "Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine"
Locations (1):
- SI "Institute of Neurology, Psychiatry and Narcology of NAMS of Ukraine", Kharkiv, Ukraine